CLINICAL TRIAL: NCT04417673
Title: A Longitudinal Survey Study on Living With Sickle Cell Disease in the COVID-19 Pandemic
Brief Title: Living With Sickle Cell Disease in the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920125; 20-HG-N125
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04-09

CONDITIONS: Isolation; Anxiety; Health Care Utilization; Sickle Cell Disease; Pain
Keywords: Mental Health; Quality of Life; Sickle Cell Pandemic Wellness; Natural History
MeSH Terms: conditions — Anxiety Disorders; Patient Acceptance of Health Care; Anemia, Sickle Cell; Pain; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Disease: Individuals with sickle cell disease

SUMMARY:
Background:

Sickle cell disease (SCD) is a chronic illness. It affects about 100,000 people in the United States. People with SCD have red blood cells that are sickle-shaped and impaired in their function. This results in a lifetime of complications that affect every organ system. People with SCD also are at greater risk for respiratory infections and lung problems. Researchers want to study how this population s stress, anxiety, fear, pain, sleep, and health care use are being affected by the COVID-19 pandemic.

Objective:

To study the extent and impact of life changes induced by the COVID-19 pandemic on people living with SCD in the U.S.

Eligibility:

People age 18 and older with SCD who live in the U.S.

Design:

Participants will complete a survey online. The questions will focus on the following:

Medical history

Mental and physical health

Demographics

Stress

Resilience

Health care use

COVID-19

Beliefs about medical mistrust and participation in research.

At the end of the survey, participants will be asked if they would like to take the survey again in the future. If they reply "yes," then they will be contacted by the study team in 6-9 months to take the survey again. They may complete the survey again in 6-8 months, 12-15 months, and 18-21 months.

The survey should take less than 40 minutes to complete.

Participants' data will be coded to protect their privacy. The coded data may be shared with other researchers.

DETAILED DESCRIPTION:
Study Description:

Longitudinal online survey of adults living with sickle cell disease (SCD) in the United States. The objective of the study is to examine the extent and impact of life changes induced by the COVID-19 pandemic on individuals living with SCD. It is our hypotheses that adults living with SCD will be adversely impacted by COVID-19 in terms of stress, anxiety, coping and sleep. Individuals living with SCD will have higher fear, isolation, anxiety and stress if they have higher clinical severity. In-person healthcare utilization for individuals with SCD will be reduced during the COVID-19 pandemic. Virtual healthcare utilization will increase for SCD individuals but satisfaction with healthcare quality will decrease.

Objectives:

Primary Objective: The primary objective of the study is to examine the extent and impact of life changes induced by the COVID-19 pandemic on individuals living with sickle cell disease (SCD). These objectives are: (1) To assess how the COVID-19 pandemic affects the psychological well-being of individuals living with SCD; (2) To examine the association between clinical severity of SCD and an individual s response to the COVID-19 pandemic; (3) To investigate whether news and other media consumption during the COVID-19 pandemic influence individual psychological well-being; (4) To determine the extent of COVID-19 induced trauma in individuals living with SCD, and its effect on health behaviors and psychological well-being; (5) To investigate the impact of the COVID-19 pandemic on healthcare utilization for SCD individuals.

Secondary Objectives: Our secondary objectives broadly examine the attitudes and viewpoints of individuals with SCD on issues of trust and the future of medical advancements for COVID-19 treatment(s). These will be examined in conjunction with the primary objectives and are: (1) To examine the role that medical and government mistrust may have on the experiences and behaviors of individuals with SCD during the pandemic; (2) To assess community attitudes towards clinical trials for COVID-19.

Endpoints:

The endpoints for the study are divided into psychosocial measures as well as physical measures and are: (1) Stress; (2) Anxiety; (3) Depressive symptomology; (4) Sleep; (5) Pain episodes and clinical severity; (6) Healthcare utilization (primary care, emergency

department, telemedicine, other). The secondary endpoint is an examination of the receptivity of SCD individuals to future health recommendations and medical treatment(s).

Study Population: Sample up to 1000 adults living with SCD in the United States, 18 years of age or older.

Description of Sites/Facilities Enrolling Participants:

Two cohorts will be recruited for this study: (1) Participants in the INSIGHTS study (NCT02156102) (2) Participants recruited by Sickle Cell 101 and/or from the NIH Study (NCT01633021), and/or from other advocacy groups or doctor s offices. Sickle Cell 101 (SC101) is a Silicon Valley-based non-profit organization that specializes in sickle cell education for the patients, caregivers, healthcare professionals, and other key stakeholders affected by sickle cell disease and trait globally.

Study Duration: Proposed enrollment opening June 1, 2020 - proposed end of data analyses from fourth wave of the study June 2022.

Participant Duration: Each participant will be invited to take the online survey every six-nine months for four data collection periods. Each survey will last 30-45 minutes.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Adults, aged 18 years or older, of any race, sex, gender, ethnicity, and/or nationality
3. Sickle Cell Disease, any genotype
4. Current Resident of the United States

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Minors less than 18 years of age
2. Adults with Sickle Cell Trait, Beta Thalassemia, Alpha Thalassemia or any blood disorder other than Sickle Cell Disorder
3. Adults who lack access to the Internet
4. Live outside the United States (unless they are from the INSIGHTS Study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Utilizing social media to reach across all scd populations in the united states.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Stress | BASELINE, MONTH 6, MONTH 12, MONTH 18
  We will examine how the COVID-19 pandemic impacts stress levels among individuals with sickle cell disease (SCD).
Pain episodes, and severity | BASELINE, MONTH 6, MONTH 12, MONTH 18
  We will examine the association between clinical severity of SCD and an individual s response to the COVID-19 pandemic.
Healthcare utilization (primary care, emergency department, telehealth other) | BASELINE, MONTH 6, MONTH 12, MONTH 18
  We will investigate the impact of the COVID-19 pandemic on healthcare utilization for SCD individuals.
Depressive symptomology | BASELINE, MONTH 6, MONTH 12, MONTH 18
  This is an examination of questions relating to depression, which we will examine within our cohort.
Anxiety | BASELINE, MONTH 6, MONTH 12, MONTH 18
  We will examine how the COVID-19 pandemic impacts anxiety levels among individuals with SCD.

SECONDARY OUTCOMES:
Receptivity to future health recommendations and medical treatment(s). | Baseline, month 6, month 12, month 18
  We would like to explore how the attitudes about treatment and levels of trust will serve as mediating factors for the experiences of individuals with SCD during this pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley J Buscetta, C.R.N.P., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hussain FA, Njoku FU, Saraf SL, Molokie RE, Gordeuk VR, Han J. COVID-19 infection in patients with sickle cell disease. Br J Haematol. 2020 Jun;189(5):851-852. doi: 10.1111/bjh.16734. Epub 2020 May 8. No abstract available. PMID 32314798